CLINICAL TRIAL: NCT03449836
Title: Effects of the Direct Interaction Between Streptococcus Salivarius 24SMBc and Streptococcus Oralis 89a With the Respiratory Epithelium in Children Affected by Allergic Rhinoconjunctivitis
Brief Title: Effects of the Direct Interaction Between Streptococcus Salivarius 24SMBc and Streptococcus Oralis 89a and the Respiratory Epithelium in Children
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Roberto Berni Canani, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 274/17
Record Dates: First submitted 2018-01-25; First posted 2018-02-28 (Actual); Last update posted 2018-03-01 (Actual); Status verified 2018-02

CONDITIONS: Allergy
MeSH Terms: conditions — Hypersensitivity | interventions — Fluticasone; Mometasone Furoate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Streptococcus salivarius 24SMBc + Strept.oralis 89a (Experimental): spray with Streptococcus salivarius 24SMBc + Strept. oralis 89a
  Interventions: Combination Product: Streptococcus salivarius 24SMBc + Strept. oralis 89a
- fluticasone + mometasone (Active Comparator): spray with fluticasone and mometasone
  Interventions: Combination Product: fluticasone + mometasone
- placebo (Placebo Comparator): spray with isotonic solution
  Interventions: Other: placebo

INTERVENTIONS:
Combination Product: Streptococcus salivarius 24SMBc + Strept. oralis 89a — nasal spray based on Streptococcus salivarius 24SMBc + Strept. oralis 89a
  Arms: Streptococcus salivarius 24SMBc + Strept.oralis 89a
Combination Product: fluticasone + mometasone — nasal spray based on fluticasone + mometasone
  Arms: fluticasone + mometasone
Other: placebo — nasal spray based on isotonic solution
  Arms: placebo

SUMMARY:
Allergic rhinoconjunctivitis is a pathology of the nasal and conjunctival mucosa induced by Immunoglobulin E (IgE) mediated inflammation following allergic exposure. This condition represents a global health problem that affects 5 to 20% of the population. As with all allergic diseases, its prevalence in pediatric age has increased over the last 30 years, as shown by the results of the international epidemiological study International Study of Asthma and Allergies in Childhood (ISAAC) which shows that the overall prevalence is 8.5 % in children aged 6-7 and 14.6% in children aged 13-14. In Italy, on average, the prevalence stands at 17.6% in the 6-7 year age range and 31.3% in the 13-14 age range, demonstrating a growing trend. The allergic rhinoconjunctivitis undiagnosed and / or not treated properly can negatively affect the school activities and in general the quality of life of children and their parents, as well as having important socio-economic repercussions in terms of medical expenses, school absences and days of work lost by parents. Furthermore, the lack of therapeutic intervention can lead to an increased risk of complications in the medium and long term. Recent advances in the understanding of the mechanisms underlying the inflammation of the airways have led to an improvement of the therapeutic strategies for the management of allergic rhinoconjunctivitis: the four cornerstones of the approach to this pathology promoted by the European Academy of Allergy and Clinical Immunology (EAACI) include allergen removal, patient education, pharmacotherapy and specific immunotherapy. However, there is discordant evidence to support their efficacy in reducing the symptomatology of allergic rhinoconjunctivitis, with the need to resort to the invasive surgical approach in several cases. Therefore, the use of probiotics, defined as "live micro-organisms which, when administered in adequate quantities, confer an advantage for the organism" can be useful. The mechanisms by which probiotics or their components, for example DNA, proteins and peptides, exert such beneficial effects concern the regulation of the immune system, the antagonist action against potentially pathogenic microorganisms and the quantitative and qualitative modulation of the intestinal microbiota. In fact, recent clinical studies have demonstrated the protective effect of infections of the high respiratory tract in adults and recurrent average otitis in pediatric age of the Streptococcus salivarius 24SMBc and Streptococcus oralis 89a strains administered through nasal spray. These well-characterized probiotics were safe, tolerated and able to positively modulate the composition of the respiratory epithelial microbiota and the function of the immune system.

ELIGIBILITY:
Inclusion Criteria:

* children aged 6-12 months with allergic rhinoconjunctivitis

Exclusion Criteria:

* concomitant presence of chronic pathologies,
* malformations of the respiratory tract and facial cranium,
* tumors,
* neurological diseases,
* metabolic pathologies,
* cystic fibrosis,
* immunodeficiencies,
* history of epistaxis,
* alteration of coagulation factors,
* history of apnea,
* ciliary dyskinesia,
* treatment with topical drugs nasal steroids and / or oral anti-histaminics or antibiotic treatment in the 3 months prior to enrollment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2018-03-01 (Estimated); Primary Completion 2018-09-30 (Estimated); Study Completion 2018-12-31 (Estimated)

PRIMARY OUTCOMES:
Total 5 Symptom Score (T5SS) from 0 to 15 | after 20 days of treatment
  Symptoms evaluation was made by the Total 5 Symptoms Score (T5SS), which includes the symptoms of nasal discharge (rhinorrhea), nasal congestion, itchy nose, sneezing, and itchy eyes. All symptoms were graded from 0 (absent) to 3 (very troublesome),with total scores ranging from 0-15.
Pittsburgh Sleep Quality Index (PSQI) score | after 20 days of treatment
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. Consisting of 19 items, the PSQI measures several different aspects of sleep, offering seven component scores and one composite score. The component scores consist of subjective sleep quality, sleep latency (i.e., how long it takes to fall asleep), sleep duration, habitual sleep efficiency (i.e., the percentage of time in bed that one is asleep), sleep disturbances, use of sleeping medication, and daytime dysfunction.
  Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the 7 component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.Traditionally, the items from the PSQI have been summed to create a total score to measure overall sleep quality.

SECONDARY OUTCOMES:
Evaluation of nasal microbiota composition | after 20 days of treatment
  Evaluation of nasal microbiota composition with a nasal brushing and determination of phyla, class, order, family, genus